CLINICAL TRIAL: NCT07352722
Title: Effect of Intercostal Mobilization on Respiratory Muscle Strength, Respiratory Function Parameters and Shuttle Walking Test Performance: A Randomized Controlled Study
Brief Title: Intercostal Mobilization and Respiratory Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Sezen Tezcan, Assist. Prof, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AIBU-FTR-ST-07
Record Dates: First submitted 2025-12-03; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intercostal Mobilization Group (Experimental)
  Interventions: Procedure: Intercostal mobilization
- Sham Group (Sham Comparator)
  Interventions: Procedure: Sham intercostal mobilization
- Control Group (Placebo Comparator)
  Interventions: Other: Rest

INTERVENTIONS:
Procedure: Intercostal mobilization — Participants lie supine, with the physical therapist performing the mobilization standing beside the bed on the side to be mobilized. For the upper ribs (ribs 1-5), the ulnar edge of the caudal hand stabilizes the upper edge of the rib below the intercostal space from the anterior side. The cranial hand grasps the participant's elbow, which is in 90° flexion of the shoulder and elbow. For the lower ribs (6th-10th ribs), the caudal hand stabilizes the upper edge of the rib below the intercostal space to be stretched anterolaterally, using the thumb and index finger to grasp the rib. Using the cranial hand, grasp the elbow at the epicondyle level and secure the participant's forearm between your own forearm and thorax. Mobilization is performed by increasing the distance between the fixation hand (caudal hand) and the mobilization hand (cranial hand). The application will be performed bilaterally with 8-10 repetitions for each intercostal space.
  Arms: Intercostal Mobilization Group
Procedure: Sham intercostal mobilization — Participants lie supine, with the physical therapist performing the mobilization standing beside the bed on the side where the mobilization will be performed. For intercostal mobilization, caudal fixation will not be performed clearly, and instead of fixing the upper edge of the rib, the caudal hand will be positioned on top of the rib. The level of distraction performed by the cranial hand will be reduced so that there is no opening in the intercostal space, and gentle stretches will be applied.
  Arms: Sham Group
Other: Rest — Individuals in the control group will be instructed to rest in a supine position for 10 minutes.
  Arms: Control Group

SUMMARY:
This cross-sectional study was planned to investigate the effects of intercostal mobilization on respiratory muscle strength, pulmonary function parameters, and performance in the ascending speed shuttle walking test. The study will be conducted in a prospective, randomized, controlled and double-blind design. A total of 90 healthy volunteers aged between 18-30 years with a sedentary lifestyle will be included in the study. The individuals will be divided into 3 groups as Intercostal Mobilization Group (n=30), Sham Application Group (n=30) and Control Group (n=30) by simple randomization. Sociodemographic Data Form, Sedentary Behavior Questionnaire, Pulmonary Function Test, Respiratory Muscle Strength Measurement (MIP/MEP), Incremental Shuttle Walking Test will be applied to the individuals before the intervention. After the intervention, only pulmonary function tests, respiratory muscle strength measurement and ISWT will be repeated. The study results are expected to contribute to the development of new evidence-based approaches to respiratory rehabilitation

DETAILED DESCRIPTION:
Breathing is one of the most fundamental biological functions that sustain life. The intake of oxygen and the expulsion of carbon dioxide are essential for sustaining life. Today, respiratory system diseases are among the major health problems worldwide, and according to World Health Organization (WHO) data, they are expected to be the third leading cause of death by 2030. Typical symptoms of these diseases include shortness of breath, coughing, depression/anxiety, fatigue, and pain. The intercostal muscles, which are among the muscles that assist in breathing, are located in the spaces between the ribs and play an important role in the expansion and contraction of the chest cavity. The external intercostal muscles are active during inspiration, while the internal intercostal muscles are active during expiration. The optimal strength and flexibility of these muscles directly affect the efficiency of lung ventilation. Osteopathic manual therapy (OMT) is a treatment approach based on the holistic relationship between body structure and function, aiming to increase structural mobility through various manual techniques. The American Osteopathic Academy describes OMT as a series of techniques focused on the principle that body structure and function are interdependent. Although OMT is not yet included among the standard treatment approaches for respiratory system diseases, it is gaining increasing attention as a complementary method to support thoracic mobility and lung function (intervertebral joints, costovertebral joints, bone structure, all ligaments, muscles, and fascia). The literature reports that applications targeting the intercostal region have positive effects such as an increase in tidal volume, improvement in chest expansion, and a decrease in dyspnea levels. Furthermore, it is stated that increased muscle activity in the intercostal muscles may lead to improvements in respiratory volume and capacity. However, the number of randomized controlled trials designed to attribute these effects solely to intercostal mobilization and conducted on young, healthy individuals is quite limited. This study aims to evaluate the effects of intercostal mobilization applications on respiratory muscle strength, respiratory function parameters, and performance in the increased-rate shuttle run test. Conducted using a randomized controlled design, this research aims to contribute to the development of evidence-based new approaches to respiratory rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 30 years old,
* Have a sedentary lifestyle,
* Be willing to participate in the study

Exclusion Criteria:

* History of neurological, orthopedic, or cardiopulmonary disease that could affect respiratory function,
* Refusal to participate in the study

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Forced expiratory volume in the first second (FEV1) | through study completion, an average of 18 months
  Forced expiratory volume in the first second (FEV1) will be assessed using a spirometer (MIR Spirobank Oxi) according to ATS and ERS criteria. The test will be repeated at least three times with forced expiration maneuvers in a sitting position, and the best value will be recorded.
Forced vital capacity (FVC) | through study completion, an average of 18 months
  Forced vital capacity (FVC) will be assessed using a spirometer (MIR Spirobank Oxi) according to ATS and ERS criteria. The test will be repeated at least three times with forced expiration maneuvers in a sitting position, and the best value will be recorded.
FEV1/FVC ratio | through study completion, an average of 18 months
  FEV1/FVC ratio will be assessed using a spirometer (MIR Spirobank Oxi) according to ATS and ERS criteria. The test will be repeated at least three times with forced expiration maneuvers in a sitting position, and the best value will be recorded.
Mid-expiratory flow rate (FEF25-75) | through study completion, an average of 18 months
  Mid-expiratory flow rate (FEF25-75) will be assessed using a spirometer (MIR Spirobank Oxi) according to ATS and ERS criteria. The test will be repeated at least three times with forced expiration maneuvers in a sitting position, and the best value will be recorded.
Peak expiratory flow (PEF) | through study completion, an average of 18 months
  Peak expiratory flow (PEF) will be assessed using a spirometer (MIR Spirobank Oxi) according to ATS and ERS criteria. The test will be repeated at least three times with forced expiration maneuvers in a sitting position, and the best value will be recorded.

SECONDARY OUTCOMES:
Respiratory muscle strength | through study completion, an average of 18 months
  Respiratory muscle strength will be assessed with a portable electronic mouth pressure device (MEC Pocket-Spiro® MPM 100) in accordance with European Respiratory Society (ERS) and American Thoracic Society (ATS) guidelines (ATS, 2002). Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using Müller and Valsalva maneuvers. For MIP, participants will exhale maximally to residual volume, then inhale rapidly to total lung capacity; for MEP, they will inhale maximally to total lung capacity and then exhale forcefully. Assessments will be performed in an upright sitting position with a nose clip, and participants will be verbally encouraged. The highest value will be recorded, provided the difference between two trials does not exceed 5% or 5 cmH₂O. Percent predicted values adjusted for age and sex will also be used
Shuttle Walking Test | through study completion, an average of 18 months
  The shuttle run test is a maximal exercise test used to evaluate aerobic capacity and functional exercise tolerance. It is performed with two cones placed 9 meters apart, creating a 10-meter course including turns. Participants walk or run back and forth in time with audio cues, starting at a low speed that increases every minute. The test ends if the participant fails to reach the cone within 0.5 meters on two consecutive cues or develops limiting symptoms (e.g., chest pain, confusion, dizziness, severe fatigue, intolerable dyspnea, SpO₂ <80%). The test consists of 12 levels and is completed when the individual reaches the maximum level or cannot continue."

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Tezcan, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No